CLINICAL TRIAL: NCT04051840
Title: Safely and Efficacy of ClinOleic-based Lipid Parenteral Nutrition After Pancreatectomy:a Prospective Study of Real World Clinical Research in China
Brief Title: Safely and Efficacy of ClinOleic-based Lipid Parenteral Nutrition
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-SR-101
Record Dates: First submitted 2019-07-31; First posted 2019-08-09 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Nutritional Supplement Toxicity
MeSH Terms: interventions — ClinOleic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ClinOleic group (Experimental): Patients will be grouped to ClinOleic-based lipid parenteral nutrition regimen using ClinOleic or Structolipid-based lipid parenteral nutrition regimen using Structolipid. From day 0 to day 5, patients will not to receive any food or liquid oral or enteral nutrition. The goal of treatment is to deliver 25kcal/kg/day, 1.05g/kg/day amino acids, and 1.1g/kg/day lipid. The weight of patient calculated as ideal body weight. The patients will be allowed water based on the clinical judgment of the Investigator. From day 6 through the remainder of the study treatment period, liquid oral or enteral nutrition could be added to the study treatment. The intent is to supply the total calculated daily nutritional requirement with study treatment plus liquid oral or enteral nutrition. Liquid oral or enteral nutrition will be increased daily, as tolerated by the patient, with a concurrent reduction in study treatment, while still supplying the calculated daily nutritional requirement.
  Interventions: Drug: ClinOleic (Baxter Healthcare, Deerfield, IL, USA)

INTERVENTIONS:
Drug: ClinOleic (Baxter Healthcare, Deerfield, IL, USA) — ClinOleic group: Patients using ClinOleic or Structolipid-based lipid parenteral nutrition regimen. From day 0 to day 5, the goal of treatment is to deliver 25kcal/kg/day, 1.05g/kg/day amino acids, and 1.1g/kg/day lipid.

SUMMARY:
Small studies suggest differences in efficacy and safety exist between olive oil-based and soybean oil-based parenteral nutrition regimens in hospitalized adult patients. A study in China suggested that olive oil-based parenteral nutrition provided effective nutrition, was well tolerated, was associated with fewer infections and conferred greater ease-of-use than soybean oil-based parenteral nutrition. The objectives of this study were to assess safety and efficacy of an ClinOleic-based lipid parenteral nutrition regimen compared with Structolipid-based lipid parenteral nutrition regimen in Chinese adults after pancreatectomy for whom oral or enteral nutrition was not possible, insufficient or contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized ≤14 days before enrolment
* required parenteral nutrition
* had the capability to complete at least five days of study treatment;
* useable peripheral vein for parenteral nutrition;
* written informed consent.

Exclusion Criteria:

* A life expectancy of <6 days;
* hypersensitivity to the study treatments;
* use of prohibited medications within 30 days before enrolment;
* serious clinically significant condition such as congestive heart failure or severe renal insufficiency;
* impaired hepatic function；
* history of human immunodeficiency virus infection;
* congenital abnormalities of amino acid metabolism;
* severe dyslipidemia;
* clinically significant abnormalities of plasma electrolytes;
* currently pregnant or lactating; prior enrolment in this clinical trial;
* participation in a clinical trial of any investigational drug or device concomitantly or within 30 days before enrolment in this clinical trial;
* unsuitable in the opinion of the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
biomarkers of liver functions | 48 hours after operation.
  Concentration of AST, ALT, TBIL, DBIL in the blood

SECONDARY OUTCOMES:
markers of infection and inflammation | 48 hours after operation.
  Concentration of CRP, PCT in the blood
Trenal function | 48 hours after operation.
  Concentration of Crea, Urea in the blood
lipids and lipid upper derivatives | 48 hours after operation.
  Concentration of arachidonic acid, eicosapentaenoic acid, linoleic acid, oleic acid in the blood

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China